CLINICAL TRIAL: NCT05075148
Title: Aneurysmal Bone Cyst Imaging After Interventional Radiology Treatment: Clinical and Radiological Outcome
Brief Title: Aneurysmal Bone Cyst Imaging After Interventional Radiology Treatment
Acronym: KOA-RI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0029
Record Dates: First submitted 2021-07-05; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-07

CONDITIONS: Bone Cysts
Keywords: Radiology, Interventional; Epidemiology; Vascualr embolisation; Percutaneous alcoholization; Aneurysmal bone cyst
MeSH Terms: conditions — Bone Cysts; Bone Cysts, Aneurysmal | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aneurysmal bone cyst: Patient aging from 0 to 30 years with diagnosis of aneurysmal bone cyst treated by percutaneous alcolisation or endovascular embolization.
  Interventions: Other: radiology

INTERVENTIONS:
Other: radiology — Interventional radiology for aneurysmal bone cyst ( percutaneous alcoholization, vascualr embolisation)

SUMMARY:
This study aims to describe the clinical outcomeand the radiological appearance of aneurysmal bone cyst treated by means of interventional radiology procedures (percutaneous sclerosis and endovascular embolization)

ELIGIBILITY:
Inclusion criteria:

* Male of female
* Aging from 0 to 30 years
* With typical aneurysmal bone cyst at initial imaging
* At least one interventional radiology procedure performed

Exclusion criteria:

* No initial surgery
* Patient refuses to participate

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Aneurysmal bone cyst
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference of size lesion after treatement | day 1
  Percentage of peripheral reossification after treatment :
  * 0%: no reossification
  * < 25%: low reossification
  * Between 25% -50%: Partial reossification
  * Between 50-75%: significant reossification
  * > 75%: very significant reossification
  * 100%: complete reossifcation

SECONDARY OUTCOMES:
Number of pain | day 1
  Pain measured with Pain scale ( 0 = no pain , 10 = maximum pain)
number of deficience | day 1
  Number of patients needs second treatment 3- Fracture ? (yes or no)
number of complication | day 1
  Fracture ? (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CYTEVAL, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC